CLINICAL TRIAL: NCT04666064
Title: Validation of COVILUS Score in Patients Suspected of COVID-19 Infection in the Emergency Room
Acronym: COVILUS2
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2020_843_0129
Record Dates: First submitted 2020-12-11; First posted 2020-12-14 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Covid19; Lung Ultrasound; Respiratory Complication
Keywords: Covid19; lung ultrasound; Respiratory Complication; triage
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Nucleic Acid Testing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Covid19 RT-PCR — patients admitted to ER for suspicion of COVID-19 infection will have a SARS-CoV-2 RT-PCR test
Other: lung ultrasound — patients admitted to ER for suspicion of COVID-19 infection who has a SARS-CoV-2 RT-PCR test and for whom the emergency doctor decide to perform a lung ultrasound

SUMMARY:
Covid-19 (English acronym meaning coronavirus disease 2019) is an emerging infectious disease caused by a strain of coronavirus called SARS-CoV-2. The current pandemic has resulted in a significant number of admissions in the emergency room (ER) due to suspicion of COVID-19 infection. Use of lung ultrasound is standard practice to diagnose acute respiratory failure in ER. Recently, typical lung ultrasonographic characteristics of COVID-19 disease has been described. The investigators demonstrated that the association of 4 signs in pulmonary ultrasound associated with a clinical sign (COVILUS score) could predict the occurrence of a positive RT-PCR in patients suspected of COVID-19 infection admitted to the emergency room. The investigators are going to conduct a new study to validate this COVILUS score in this type of patient. The main objective will be to validate the diagnostic performance of lung ultrasound in patients admitted to the emergency room with suspected COVID19 infection.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to ER for suspicion of COVID-19 infection who has a SARS-CoV-2 RT-PCR test and for whom the emergency doctor decide to perform a lung ultrasound as part of the BLUE protocol
* Age> 18 years old

Exclusion Criteria:

* patients < 18 years of age
* patients under guardianship or curators
* pregnancy
* poor echogenicity due to the presence of an acoustic barrier (pneumothorax, subcutaneous emphysema, etc.)
* patients with a suspected or proven acute lung disease (pneumonitis, acute respiratory distress syndrome (ARDS))
* patients with chronic interstitial lung disease
* patients who will refuse to give their consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted to ER for suspicion of COVID-19 infection who has a SARS-CoV-2 RT-PCR test and for whom the emergency doctor decide to perform a lung ultrasound as part of the BLUE protocol
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-04-28 (Actual)

PRIMARY OUTCOMES:
concordance between Covid19 RT-PCR results and lung ultrasound results | one week

CONTACTS AND LOCATIONS:
Locations (1):
- BAR, Amiens, France

IPD SHARING:
Plan to Share IPD: No